CLINICAL TRIAL: NCT00002128
Title: Phase I Study of the Safety, Tolerance, and Pharmacokinetics of 9-[2-(Bispivaloyloxymethyl)Phosphonylmethoxyethyl]Adenine (Bis-POM PMEA; Adefovir Dipivoxil) in HIV-Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 232A; GS-93-401
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1994-07

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents; Adenine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — adefovir dipivoxil

INTERVENTIONS:
Drug: Adefovir dipivoxil

SUMMARY:
To study the safety, tolerance, and pharmacokinetics of a single dose of bis-POM PMEA (adefovir dipivoxil) when administered by the oral route in patients with HIV infection.

DETAILED DESCRIPTION:
Five patients are entered at each of three dose levels of bis-POM PMEA administered orally in a single dose.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* AZT, ddI, or ddC (provided patient has been on a stable regimen for at least 4 weeks prior to study entry).
* Prophylactic aerosolized pentamidine, fluconazole, ketoconazole, trimethoprim/sulfamethoxazole, or dapsone (provided patient has been on a stable regimen for at least 4 weeks prior to study entry).

Patients must have:

* Documented HIV infection or diagnosis of AIDS.
* Life expectancy of at least 3 months.

Prior Medication:

Allowed:

* Prior AZT, ddI, or ddC.
* Prophylactic aerosolized pentamidine, fluconazole, ketoconazole, trimethoprim/sulfamethoxazole, or dapsone.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Active, serious infections (other than HIV infections) that require parenteral antibiotic therapy.
* Clinically significant cardiac disease, including symptoms of ischemia, congestive heart failure, or arrhythmia.
* Gastrointestinal malabsorption syndrome or inability to receive oral medication.

Concurrent Medication:

Excluded:

* Diuretics.
* Amphotericin B.
* Aminoglycoside antibiotics.
* Parenteral antibiotics.
* Other nephrotoxic agents.
* Other investigational agents.
* Non-steroidal anti-inflammatory drugs.
* Aspirin.

Prior Medication:

Excluded within 2 weeks prior to study entry:

* Diuretics.
* Amphotericin B.
* Aminoglycoside antibiotics.
* Parenteral antibiotics.
* Other nephrotoxic agents.
* Other investigational agents.

Excluded within 3 days prior to study entry:

* Non-steroidal anti-inflammatory drugs.
* Aspirin. Active substance abuse (including alcohol or drug abuse).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Univ, Baltimore, Maryland, United States

REFERENCES:
- [Background] Cundy KC, Barditch-Crovo P, Walker RE, Collier AC, Ebeling D, Toole J, Jaffe HS. Clinical pharmacokinetics of adefovir in human immunodeficiency virus type 1-infected patients. Antimicrob Agents Chemother. 1995 Nov;39(11):2401-5. doi: 10.1128/AAC.39.11.2401. PMID 8585716